CLINICAL TRIAL: NCT00317031
Title: Individually Adapted Therapy of Alcoholism: Clinical Studies
Brief Title: Individually Adapted Therapy of Alcoholism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Merck Sharp & Dohme LLC (Industry); Dupont Applied Biosciences (Industry)
Responsible Party: Kiefer, Falk, Central Institute of Mental Health (CIMH), Mannheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PREDICT
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Alcoholism
Keywords: Alcoholism; Drug Therapy
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- 1 (Active Comparator): Acamprosate
  Interventions: Drug: Acamprosate or Naltrexone
- 2 (Active Comparator): Naltrexone
  Interventions: Drug: Acamprosate or Naltrexone
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Acamprosate or Naltrexone

INTERVENTIONS:
Drug: Acamprosate or Naltrexone — mg&d 90 days

SUMMARY:
The primary objective is to directly compare the efficacy of acamprosate, naltrexone and placebo for relapse prevention in alcoholics.

DETAILED DESCRIPTION:
The primary objective is to directly compare the efficacy of acamprosate, naltrexone and placebo for relapse prevention in alcoholics. The secondary objective is to establish an association between patients' motivational type and drug effects. The aim is to improve alcoholism treatment by identifying characteristics for response to specific pharmacological relapse prevention. Such items could allow for an individually adapted pharmacotherapy of alcoholism. Specifically, we will study the possible dependence of the efficacy of naltrexone and/or acamprosate on different motivational types (reward versus relief craving) and genetic profiles referring to glutamatergic and opioidergic candidate genes. Lastly, the longterm costs and cost-effectiveness of the different treatment strategies for alcoholics chosen in our study are established.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will have a current DSM-IV/ICD 10 diagnosis of alcohol dependence.
2. Participants must have had a minimum of 14 drinks (females) or 21 drinks (males) on average per week over a consecutive 30-day period in the 90-day period prior to initiation of abstinence, and must have had two or more days of heavy drinking (defined as 4 drinks for females and 5 drinks for males) in the 90-day period prior to initiation of abstinence.
3. Participants must have had a minimum of 72 hours of abstinence and no significant withdrawal symptoms (CIWA < 8) prior to randomization.
4. At least 2 weeks of inpatient treatment.
5. Participants can be abstinent for a maximum of 28 days prior to randomization.
6. Participants are willing not to seek additional psychotherapy during the first 6 months of study except attendance of mutual help groups.
7. Participants have to sign a witnessed declaration of informed consent.

Exclusion Criteria:

1. Participants who meet current DSM-IV criteria for bipolar disorder, schizophrenia, bulimia/anorexia, dementia, or a psychological disorder for whom medication is indicated, but no other Axis I disorders that are not medicated and are not severe enough to require medications.
2. Participants who require psychopharmacotherapy.
3. Participants who require therapy with any medications which pose safety issues.
4. Participants with a current abuse of any psychoactive drug and who show a positive drug test on an urine screen.
5. Participants with a lifetime diagnosis of dependence on any psycho-active drug except for nicotine or habitual caffeine use.
6. Participants who have significant medical disorders which would increase the potential risk of the study treatment or interfere with the study participation.
7. Participants with abnormal AST or ALT (more than 5 times the normal level).
8. Participants who are pregnant or nursing infant(s).
9. Women during childbearing years without an effective contraceptive method.
10. Participants developing sensitivity to the study medication.
11. Participants who are illiterate or are unable to read and write German.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2002-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
time to relapse to heavy drinking (consumption of more than 48 gram alcohol/day for females and more than 60 gram alcohol/day for males) | 06/2008

SECONDARY OUTCOMES:
percentage of days without heavy drinking (consumption of more than 48 gram alcohol/day for females and more than 60 gram alcohol/day for males) | 06/2008
time to first alcohol consumption | 06/2008
percentage of days of complete abstinence from alcohol | 06/2008

CONTACTS AND LOCATIONS:
Overall Officials: Karl F. Mann, MD, Principal Investigator — Central Institute of Mental Health, J5, 68159 Mannheim, Germany; Michael N. Smolka, MD, Principal Investigator — Central Insitute of Mental Health, J5, 68159 Mannheim, Germany
Locations (5):
- Germany (5):
  - Department of Psychiatry, University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Department of Psychiatry, University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - Department of Addictive Behavior und Addiction Medicine, Central Institute of Mental Health, Mannheim, Baden-Wurttemberg
  - Department of Psychiatry, University of Tübingen, Tübingen, Baden-Wurttemberg
  - Department of Psychiatry, University of Regensburg, Regensburg, Bavaria

REFERENCES:
- [Derived] Reinhard I, Lemenager T, Fauth-Buhler M, Hermann D, Hoffmann S, Heinz A, Kiefer F, Smolka MN, Wellek S, Mann K, Vollstadt-Klein S. A comparison of region-of-interest measures for extracting whole brain data using survival analysis in alcoholism as an example. J Neurosci Methods. 2015 Mar 15;242:58-64. doi: 10.1016/j.jneumeth.2015.01.001. Epub 2015 Jan 12. PMID 25593047
- [Derived] Mann K, Vollstadt-Klein S, Reinhard I, Lemenager T, Fauth-Buhler M, Hermann D, Hoffmann S, Zimmermann US, Kiefer F, Heinz A, Smolka MN. Predicting naltrexone response in alcohol-dependent patients: the contribution of functional magnetic resonance imaging. Alcohol Clin Exp Res. 2014 Nov;38(11):2754-62. doi: 10.1111/acer.12546. PMID 25421512
- [Derived] Lemenager T, Hill H, Reinhard I, Hoffmann S, Zimmermann US, Hermann D, Smolka MN, Kiefer F, Vollstadt-Klein S, Heinz A, Mann K. Association between alcohol-cue modulated startle reactions and drinking behaviour in alcohol dependent patients - results of the PREDICT study. Int J Psychophysiol. 2014 Dec;94(3):263-71. doi: 10.1016/j.ijpsycho.2014.09.009. Epub 2014 Sep 28. PMID 25269022
- [Derived] Mann K, Lemenager T, Hoffmann S, Reinhard I, Hermann D, Batra A, Berner M, Wodarz N, Heinz A, Smolka MN, Zimmermann US, Wellek S, Kiefer F, Anton RF; PREDICT Study Team. Results of a double-blind, placebo-controlled pharmacotherapy trial in alcoholism conducted in Germany and comparison with the US COMBINE study. Addict Biol. 2013 Nov;18(6):937-46. doi: 10.1111/adb.12012. Epub 2012 Dec 12. PMID 23231446